CLINICAL TRIAL: NCT05610358
Title: Efficacy of Smartphone Application Based Rehabilitations in Patients With Chronic Respiratory or Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-1460
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Rehabilitation; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will be provided the smartphone application and they will practice application based rehabilitation for 12 weeks.
  Interventions: Device: smartphone application
- Control (No Intervention): Participants in the control group will not practice rehabilitation program.

INTERVENTIONS:
Device: smartphone application — In this study, the investigators will provide smartphone application based 12-week pulmonary or cardiac rehabilitation program to patients with chronic respiratory or cardiovascular diseases.
  Arms: Intervention

SUMMARY:
In Republic of Korea, it is not easy to practice standard pulmonary rehabilitation (PR) or cardiac rehabilitation (CR). In this study, the investigators will provide newly developed smartphone application to patients with chronic respiratory or cardiovascular diseases. The investigators want to confirm whether participants, who perform smartphone application based 12-week PR or CR program, present improved exercise capacity, dyspnea symptom, muscle strength, or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea symptom >= mMRC 1 or NYHA II
* adults between 20 years and 80 or years

  * Chronic respiratory disease
* FEV1/FVC < 0.7 or FEV1< 0.8 of predicted value in pulmonary function test
* bronchiectasis in more than one lobe on chest computed tomography
* FVC or DLCO < 0.8 of predicted value in pulmonary function test

  * Chronic cardiovascular disease
* Reperfusion Therapy for angina pectoris or myocardial infarction
* Heart failure with reduced ejection fraction (LVEF < 50%)

Exclusion Criteria:

* history of acute exacerbation within 4 weeks
* unable to comply rehabilitation program
* not suitable for study on decision by duty physician
* no consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
change of maximal oxygen consumption (VO2max) | 12 weeks
  The maximal oxygen consumption (VO2max) is measured during incremental exercise test (cardiopulmonary exercise test).
Change of Chronic obstructive pulmonary disease (COPD) assessment Test (CAT) (Chronic respiratory disease group) | 12 weeks
  Self reported Patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status. Each item is scored 0-5, yielding a total between 0 and 40
change of Korean Health-related Quality of Life Instrument with 8 Items (HINT-8) score (Chronic cardiovascular disease group) | 12 weeks
  A questionnaire assessing health related quality of life on 4 health dimensions (physical, mental, social, positive health dimension). Each item is scored 1-4, yielding a total between 8 and 40.
  The scores range from 8 (best performance) to 40 (worst performance).

SECONDARY OUTCOMES:
change of dyspnea symptom (Chronic respiratory disease group) | 12 weeks
  Dyspnea symptom is measured according to the Modified Medical Research Council (mMRC) Dyspnea Scale.
  The mMRC scale is from 0 to 4:
  0: no breathlessness except on strenuous exercise
  1. shortness of breath when hurrying on the level or walking up a slight hill
  2. walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level
  3. stops for breath after walking ∼100 m or after few minutes on the level
  4. too breathless to leave the house, or breathless when dressing or undressing
change of dyspnea symptom (Chronic cardiovascular disease group) | 12 weeks
  Dyspnea symptom is measured according to the New York Heart Association Functional Classification (NYHA class).
  The NYHA class is from I to IV:
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation (feeling heart beats), or dyspnea (shortness of breath).
  Class II(Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III(Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV(Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
Change of EuroQol 5-dimension 5-level (EQ-5D-5L) score | 12 weeks
  A questionnaire assessing health related quality of life on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each item is scored 1-5, yielding a total between 5 and 25.
  The scores range from 5 (best performance) to 25 (worst performance).
change of Korean Health-related Quality of Life Instrument with 8 Items (HINT-8) score (Chronic respiratory disease group) | 12 weeks
  A questionnaire assessing health related quality of life on 4 health dimensions (physical, mental, social, positive health dimension). Each item is scored 1-4, yielding a total between 8 and 40.
  The scores range from 8 (best performance) to 40 (worst performance).
change of hand grip strength | 12 weeks
  The muscle strength measures hand grip strength. The cut-off value for sarcopenia is < 30 kg
change of limb muscle mass | 12 weeks
  The muscle mass is measured using the Bioelectrical Impedance Analysis. The cut off value for sarcopenia is < 7.26 kg/m^2.
change of forced expiratory volume in one second (FEV1) (Chronic respiratory disease group) | 12 weeks
  The forced expiratory volume in one second (FEV1) is measured using spirometry. The value will be presented in % predicted value.
change of forced vital capacity (FVC) (Chronic respiratory disease group) | 12 weeks
  The forced vital capacity (FVC) is measured using spirometry. The value will be presented in % predicted value.
change of diffusing capacity of the lung for carbon monoxide (DLCO) (Chronic respiratory disease group) | 12 weeks
  The diffusing capacity of the lung for carbon monoxide (DLCO) is measured using single breath holding method.
  The value will be presented in % predicted value.
Change of chest pain symptom (Chronic cardiovascular disease group) | 12 weeks
  Chest pain symptom is measured according to the Canadian Cardiovascular Society grading of angina pectoris (CCS angina grade).
  The CCS angina grade is from I to IV:
  Grade I: Angina with strenuous/rapid/prolonged exertion at work or recreation only; no angina with ordinary physical activity, e.g. walking, climbing stairs Grade II: Ordinary activity slightly limited: angina with walking/climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold/wind, under emotional stress, during few hours after awakening, walking >2 blocks on level ground, or climbing >1 flight of stairs at normal pace and normal conditions Grade III: Marked limitation of ordinary physical activity: angina with walking 1-2 blocks on level ground or climbing 1 flight of stairs at normal pace and normal conditions Grade IV: Inability to carry on any physical activity without discomfort; anginal syndrome may be present at rest
change of exercise duration in cardiopulmonary exercise test (Chronic cardiovascular disease group) | 12 weeks
  This test measures total exercise duration.
change of exercise capacity in cardiopulmonary exercise test (Chronic cardiovascular disease group) | 12 weeks
  This test measures metabolic equivalents (METs).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request.

REFERENCES:
- [Derived] Chung C, Kim AR, Kang DY, Kim S, Oh J, Kim HJ, Park B, Lee SH, Kim D, Kwon H, Jo MW, Lee SW. Clinical Efficacy of Smartphone App-Based Pulmonary Rehabilitation in Chronic Respiratory Diseases: Randomized Controlled and Feasibility Trials. J Med Internet Res. 2025 Nov 28;27:e76801. doi: 10.2196/76801. PMID 41313804
- [Derived] Chung C, Kim AR, Jang IY, Jo MW, Lee S, Kim D, Kwon H, Kang DY, Lee SW. Smartphone application-based rehabilitation in patients with chronic respiratory and cardiovascular diseases: a randomised controlled trial study protocol. BMJ Open. 2023 Sep 20;13(9):e072698. doi: 10.1136/bmjopen-2023-072698. PMID 37730392